CLINICAL TRIAL: NCT04935047
Title: A Feasibility Study and a Pilot Randomised Trial of a Multilingual Support Intervention to Improve Norwegian Language Skills for Refugees
Brief Title: Pilot Trial of Multilingual Support Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 914633
Record Dates: First submitted 2021-06-02; First posted 2021-06-22 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2021-05

CONDITIONS: Language
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Multilingual Support) (Experimental): The treatment group will receive seven hours multilingual support weekly.
  Interventions: Other: Multilingual Support
- Control group (No Intervention): The control group will receive the same amount of support as the experimental group, but from a person without multilingual qualifications.

INTERVENTIONS:
Other: Multilingual Support — Multilingual Support is a classroom intervention, which is designed to be delivered in classes of adult learning of a new language. The intervention involves the use of a language assistant, who is at minimum independent user (B1) in the language to be learned (in this case Norwegian), according to the language proficiency scale of the Common European Framework of Reference (CEFR) for languages, learning, teaching, assessment (Little, 2006). The language assistant will be in the classroom for seven hours a week, collaborating with the teacher in providing language training. In classrooms where participants have different primary languages, the language assistant(s) must cover all languages represented in the classroom.
  Arms: Experimental (Multilingual Support)

SUMMARY:
This is a feasibility study and a pilot trial of a multilingual support intervention with the aim to improve language training for Norwegian refugees by systematically using the participants' primary language to support the learning of the new language. The study is conducted in three Norwegian municipalities with the aim to evaluate feasibility for a full-scale randomised controlled trial. The pilot trial will include at least 30 participants, with two thirds allocated to the treatment group and one third to the control group. The intervention will be implemented as an add on to ordinary classroom settings. The treatment group will receive seven hours multilingual support weekly. The control group will receive the same amount of support, but from a person without multilingual qualifications. The Norwegian Directorate of Integration and Diversity (IMDi) are funding the project and have reviewed the protocol.

DETAILED DESCRIPTION:
Design

The pilot trial is designed as an individual randomised study in three sites, conducted from August 2021 to June 2022. Participants randomised to treatment condition will receive language training with Multilingual Support. Participants randomised to control condition will receive language training without Multilingual Support. The number of assistants in the classroom will be equal in treatment and control condition, however, only the assistants in treatment condition will master the participants' primary language and follow the guidelines set out in Multilingual Support manual.

Participants

To be eligible for participation, persons must be at early stages of their language learning (i.e. below A2 levels), and eight or less years of education in primary and lower secondary school. In order to limit the number of languages provided by the Multilingual assistants, and hence reduce the complexity of the study, we pilot the intervention and trial within the one or two largest language groups at each site (i.e. Arabic and Kinyabwisha/Swahili in pilot 1; Coastal town; Arabic and Dari in pilot 2; Middle-town; and Arabic in pilot 3; Suburb-town. Persons who are illiterate are excluded from the study.

Recruitment

Staff at the local Adult Vocational centre identify eligible participants for language training with Multilingual Support from June to August 2021. When an eligible person has been identified, the staff provides the person with information about the study. This information will be provided in writing in Norwegian and in the person's primary language. In addition, the information will be given orally, in eligible participants primary language, making it possible for eligible participants to ask questions about the project. If the person agrees to participate in the study, the staff deliver the participants email address and information about their primary language to the researchers. Only participants that provide written content will be included in the study.

Randomisation procedures

When receiving the participant's email address and information on primary language, the researchers send a request to the participant, inviting him/her to respond to a baseline survey. When responding to the baseline survey, participants are not aware of their allocation to treatment or control condition. The survey client (Nettskjema.no) includes a function to randomise participants. In this study we randomise participants into two groups, with 2/3 probability of being allocated to the treatment condition. Randomisation is conducted as independent randomisation (no stratification). After the participant has submitted the baseline survey, the researchers can obtain information on treatment allocation, and inform the staff at the local Adult Vocational centre about the randomisation result, whereafter the Centre invites the participant to the Multilingual Support or the control condition.

ELIGIBILITY:
Inclusion criteria:

* early stages of their language learning (i.e. below A2 levels), and
* eight or less years of education in primary and lower secondary school, and
* a major language equal to one of the Multilingual assistants.

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in language skills | Change from Baseline language skills at 10 months
  Language tests, administered by the Norwegian Directorate for Lifelong Learning. Scale: 0-100% correct answers. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change in Self-Efficacy in Norwegian language | Change from Baseline Self-Efficacy in Norwegian language at 8 months
  The short Norwegian version of the English Self-Efficacy Questionnaire (Wang, Kim, Bai, & Hu, 2014). Developed with a 7 point likert scale, but we apply a 5 point likert scale. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Grete G Tøge, phd, Principal Investigator — associate professor
Locations (3):
- Norway (3):
  - Ålesund VO, Ålesund
  - Drammen VO, Drammen
  - Lillestrøm VO, Lillestrøm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tøge, Anne Grete; Malmberg-Heimonen, Ira; Søholt, Susanne; Vilhjalmsdottir, Sigridur (2022). Protocol: Feasibility study and pilot randomised trial of a multilingual support intervention to improve Norwegian language skills for adult refugees. International Journal of Educational Research . Vol. 112.